CLINICAL TRIAL: NCT05537909
Title: Role of Gut Microbiota in the Pathophysiology of Aseptic Abscesses
Acronym: ABSCESSBIOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RBHP ANDRE (ABSCESSBIOT); 2017-A03499-44 (Other: ANSM)
Record Dates: First submitted 2022-06-17; First posted 2022-09-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-02

CONDITIONS: Aseptic Abscess Syndrome
Keywords: Aseptic abscess syndrome; Comparative Study; Pathophysiology

STUDY DESIGN:
Intervention Model Description: All patients and their controls will have a sample of urine, stool, saliva and blood taken during a follow-up visit. Patients will not be specifically asked to take these samples, they will be taken during a follow-up visit, during which these samples are usually already taken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Experimental): adult patients with aseptic abscess syndrome
  Interventions: Other: Biological sample collection
- control (Experimental): control An adult person living in the same environment as the case.
  Interventions: Other: Biological sample collection

INTERVENTIONS:
Other: Biological sample collection — All patients and their controls will be asked to provide a urine, stool, saliva and blood sample during a follow-up visit. Patients will not be specifically asked to take these samples, they will be taken during a follow-up visit, during which these samples are usually already taken.

SUMMARY:
Aseptic abscess syndrome (AA) is a rare entity characterized by the occurrence of deep abscesses with no germ found. Antibiotic therapy is ineffective and they are sensitive to anti-inflammatory treatment with corticosteroids.

Gut microbiota is important for the development of the immune system. In Crohn's disease which is frequently associated with AA syndrome, dysbiosis is found but could also be involved in the immune response at a distance from the gut.

Stool, blood, saliva and urine samples will be taken from the patients included and their controls in the centers where they are followed. These biological samples will be transported to Clermont Ferrand using the same procedure (transporter and dry ice) where the following analyses will be performed: microbiota on stool and saliva, short chain fatty acids on stool and lymphocyte study on blood.

DETAILED DESCRIPTION:
* Included patients will be adult patients meeting the diagnostic criteria for aseptic abscess syndrome described by André et al.
* Controls will be adults without aseptic abscess syndrome living in the same environment as the patients, whether related to the patient or not.

Patients and controls must be able to provide informed consent and be affiliated with the French Social Security system.

ELIGIBILITY:
Inclusion Criteria:

* For cases: adult patients meeting the diagnostic criteria for aseptic abscess syndrome described by André et al:
* Deep abscesses on radiological examination with neutrophilic features proven by pathological analysis of a surgical specimen or biopsy when performed
* Negative blood cultures, negative serological tests for bacteria, including always Yersinia enterocolitica, and, during surgery or aspiration, sterile pus (with standard cultures, BAAR and fungal tests) Failure of antibiotic therapy, when prescribed, after at least 2 weeks for conventional antibiotic therapy and at least 3 months for anti-tuberculosis treatment
* Rapid clinical improvement the day after the prescription of corticosteroids (at least 1/2 mg/kg prednisone or equivalent) followed by radiological improvement after 1 month of corticosteroids, sometimes in association with immunosuppressive treatments.

For controls: adult person living in the same environment as the case to which it is matched. Adult person living in the same household or near the patient.

For cases and controls:

* Ability to provide informed consent.
* Membership in the Social Security system.

Exclusion Criteria:

* Pregnant women. Incapable patients Patients deprived of liberty Antibiotic therapy administered within 6 weeks prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota profiling (diversity) of patients with aseptic abscess syndrome and matched healthy controls | day 1
  16S rRNA gene sequencing technique and illumina MiSeq platform to investigate the difference of gut microbiota composition between patients with aseptic abscess syndrome and matched healthy controls.
Gut microbiota profiling (composition) of patients with aseptic abscess syndrome and matched healthy controls | day 1
  16S rRNA gene sequencing technique and illumina MiSeq platform to investigate the difference of gut microbiota diversity between patients with aseptic abscess syndrome and matched healthy controls.

SECONDARY OUTCOMES:
Th17/Treg Lymphocytes phenotyping | day 1
  Th17/Treg Lymphocytes phenotyping of patients with aseptic abscesses compared to matched healthy controls.
Salivary microbiota profiling (composition) of patients with aseptic abscess syndrome and matched healthy controls | day 1
  16S rRNA gene sequencing technique and illumina MiSeq platform to investigate the difference of salivary microbiota composition between patients with aseptic abscess syndrome and matched healthy controls.
Salivary microbiota profiling (diversity) of patients with aseptic abscess syndrome and matched healthy controls | day 1
  16S rRNA gene sequencing technique and illumina MiSeq platform to investigate the difference of salivary microbiota diversity between patients with aseptic abscess syndrome and matched healthy controls.

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - CHU de Bordeaux, Bordeaux
  - Centre Hospitalier Intercommunal Nord-Ardennes, Charleville-Mézières
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU Henri Mondor - Assistance Publique -Hôpitaux de Paris (AP-HP), Créteil
  - Centre Hospitalier de Dax, Dax
  - Centre Hospitalier Saint Joseph Saint Luc, Lyon
  - Hospices Civils de Lyon, Lyon
  - Assistance Publique - Hôpitaux de Marseille (AP-HM), Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - CHU de Nimes, Nîmes
  - Hôpital Cochin - Assistance Publique -Hôpitaux de Paris (AP-HP), Paris
  - Hôpital La Pitié-Salpétrière - Assistance Publique -Hôpitaux de Paris (AP-HP), Paris
  - Hôpital Louis Mourier - Assistance Publique -Hôpitaux de Paris (AP-HP), Paris
  - Hôpital Saint Louis Lariboisière - Assistance Publique -Hôpitaux de Paris (AP-HP), Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trefond L, Billard E, Pereira B, Richard D, Vazeille E, Bonnet R, Barnich N, Andre M; Aseptic Abscess Syndrome physicians. Host-microbiota relationship in the pathophysiology of aseptic abscess syndrome: protocol for a multicentre case-control study (ABSCESSBIOT). BMJ Open. 2023 Aug 4;13(8):e073776. doi: 10.1136/bmjopen-2023-073776. PMID 37541750